CLINICAL TRIAL: NCT01583231
Title: Efficacy of the Brushless Scrub
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Theresa Criscitelli, Director of Perioperative Education, Winthrop University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 302192-1
Record Dates: First submitted 2012-02-21; First posted 2012-04-23 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Focus of Study: Handwashing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Prewash (No Intervention): Level 1: participants will be swabbed, then application of brushless scrub, swabbed again
- Prewash (Experimental): Level 2: participants will be swabbed, perform a wash with soap and water for 1 minute, dry, apply brushless scrub, swabbed again
  Interventions: Other: Prewash

INTERVENTIONS:
Other: Prewash — The intervention will be the addition of the prewash utilizing non-antimicrobial soap and water.
  Arms: Prewash

SUMMARY:
The aim of this research is to examine if the brushless scrub is effective in reducing bioburden on the hands of the operating room (OR) personnel both with a prewash of one minute prior to scrub and without a prewash prior to scrub, and to compare the bioburden reduction between both methods.

Hypothesis I: A soap and water prewash used prior to brushless scrub further decreases bioburden than brushless scrub alone.

Hypothesis II: Brushless scrub is effective in reducing the bioburden measured just after the application of the brushless scrub within 20 seconds of application for both groups.

Exploratory Hypothesis: We will also compare the bioburden measured before and at 1.5 minutes after application of the brushless scrub for both groups.

DETAILED DESCRIPTION:
Hand washing by operating room personnel prior to surgical procedures is essential in the prevention of intraoperative infection. The use of the brushless surgical hand hygiene has been used since the CDC stated in 2002 that using a brush and sponge is no longer necessary. Empirical literature supports the reduction of the incidence of bacteria or OR personnel hands with the use of alcohol-based products.

An annotated integrative search of the literature was conducted and conflicting information regarding the use of a prewash prior to the brushless scrub was found. This study can help us utilize the brushless scrub to the fullest capacity and prevent surgical site infections.

The time point at which the outcome measure will be assessed at an individual level will be immediately pre-intervention and also 1.5 minutes after the intervention. For example, within 15 seconds prior to brushless scrub, or prewash, a sample swab will be collected and then another sample swab will be obtained 1.5 minutes later for postintervention measure. The study should take approximately 4 months to complete to get an adequate sample size of individuals for statistical power. The data will be aggregated and presented at a staff in-service within 3 months after data collection and analysis is completed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion will consist of all OR personnel and students who scrub for surgical procedures.

Exclusion Criteria:

* Exclusion will consist of any OR personnel and students whom do not want to participate in the study or those who have not been part of the the routine and mandatory training of proper surgical hand hygiene which occurs annually.

Ages: 19 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Reduction of bioburden | 1.5 minutes after brushless scrub was applied
  The procedure of swabbing the participants will be measured by using the RUHOF ATP Complete Contamination Monitoring System.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Criscitelli, MS, RN, CNOR, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] Heeg P, Ostermeyer C, Kampf G. Comparative review of the test design Tentative Final Monograph (TFM) and EN 12791 for surgical hand disinfectants. J Hosp Infect. 2008 Oct;70 Suppl 1:22-6. doi: 10.1016/S0195-6701(08)60007-9. PMID 18994678
- [Result] Kampf G, Kramer A. Epidemiologic background of hand hygiene and evaluation of the most important agents for scrubs and rubs. Clin Microbiol Rev. 2004 Oct;17(4):863-93, table of contents. doi: 10.1128/CMR.17.4.863-893.2004. PMID 15489352
- [Result] Hubner NO, Kampf G, Kamp P, Kohlmann T, Kramer A. Does a preceding hand wash and drying time after surgical hand disinfection influence the efficacy of a propanol-based hand rub? BMC Microbiol. 2006 Jun 22;6:57. doi: 10.1186/1471-2180-6-57. PMID 16790073
- [Result] Kampf G, Ostermeyer C. A 1-minute hand wash does not impair the efficacy of a propanol-based hand rub in two consecutive surgical hand disinfection procedures. Eur J Clin Microbiol Infect Dis. 2009 Nov;28(11):1357-62. doi: 10.1007/s10096-009-0792-7. Epub 2009 Aug 11. PMID 19669812